CLINICAL TRIAL: NCT05946174
Title: Tackling Disruptions to Frailty Interventions: Developing Personalized Interventions Targeted for Older Persons With Cardiac Frailty
Acronym: INDEPENDENCY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/2086
Record Dates: First submitted 2023-06-15; First posted 2023-07-14 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Diseases
Keywords: Frailty; Intervention; Cardiac Frailty Interventions
MeSH Terms: conditions — Cardiovascular Diseases; Frailty

STUDY DESIGN:
Intervention Model Description: Set A comprises of outpatient clinic/ community participants, who will be randomized in a 1:1 ratio into Group A1 (receiving Intervention Set A- exercise sessions and meals over approximately 12 weeks) or Group A2 (control/ usual care)
  Set B comprises of step-down community hospital participants, who will be randomized in a 1:1 ratio into Group B1 (receiving Intervention Set B- exercise sessions and meals over approximately 3 weeks) or Group B2 (control/ usual care)
  Set C comprises of acute community hospital participants, who will be randomized in a 1:1 ratio into Group C1 (receiving Intervention Set C- meals over approximately 3 weeks) or Group C2 (control/ usual care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Outpatient clinic/community participants receiving exercise sessions and meals (A1) (Experimental): Outpatient clinic/community participants receiving intervention Set A (exercise sessions and meals over approximately 12 weeks)
  Interventions: Other: Intervention Set A
- Outpatient clinic/community participants receiving control/usual care (A2) (No Intervention): Outpatient clinic/community participants receiving control/usual care
- Step-down community hospital participants receiving exercise sessions and meals (B1) (Experimental): Step-down community hospital participants receiving Intervention Set B (exercise sessions and meals over approximately 3 weeks)
  Interventions: Other: Intervention Set B
- Step-down community hospital participants receiving control/usual care (B2) (No Intervention): Step-down community hospital participants receiving control/usual care
- Acute hospital participants receiving meals (C1) (Experimental): Acute hospital participants receiving Intervention Set C (meals over approximately 3 weeks)
  Interventions: Other: Intervention Set C
- Acute hospital participants receiving control/usual care (C2) (No Intervention): Acute hospital participants receiving control/usual care

INTERVENTIONS:
Other: Intervention Set A — exercise sessions and meals over approximately 12 weeks
  Arms: Outpatient clinic/community participants receiving exercise sessions and meals (A1)
Other: Intervention Set B — exercise sessions and meals over approximately 3 weeks
  Arms: Step-down community hospital participants receiving exercise sessions and meals (B1)
Other: Intervention Set C — meals over approximately 3 weeks
  Arms: Acute hospital participants receiving meals (C1)

SUMMARY:
Background: Muscle mass loss and metabolic dysfunction, exacerbated by inactivity and nutritional inadequacies, underpin both cardiovascular disease and frailty in ageing. The investigators' proposal seeks to develop interventions in exercise and diet that are targeted for older adults with cardiac frailty.

Methods:

The investigators' proposal is a five-year study comprising of first phase (first 2-2.5 years) and second phase (next 2-2.5 years). In the first phase cardiac frail participants (up to N=500) from each healthcare transition (inpatient hospital, step-down community hospital, outpatient clinic/community) will be randomized to receive Intervention Sets or usual care. The second phase will scale up these programs. Three Intervention Sets A, B, and C will be implemented in the outpatient, step-down community hospital, and acute hospital settings. Diet intervention comprises meal sets prepared with nutrients involved in energy metabolism. Exercise training is facilitated by hospital gyms and hospital physiotherapists. Diet and exercise behavior will be monitored using questionnaires, video conferencing and meal photos.

Significance: Clinical studies are urgently needed using consistent frailty tools to evaluate the efficacy and promise of frailty interventions, targeted to achieve reversal/retardation of frailty. When scaled up, these approaches will provide high-quality science needed to manage cardiac frailty towards healthier population ageing.

DETAILED DESCRIPTION:
BACKGROUND Cardiovascular disease is a formidable disruptor of interventions related to exercise intervention. Patients and physicians face uncertainty about dispensing safe and effective exercise programs to frail patients with concomitant cardiovascular disease. This hesitancy permeates across transitions from acute to step-down care to community settings. Uncertainties include fear of exacerbating heart conditions, individual variability in exercise response and what exercise targets to reach that is rational for each patient. Often, little or no exercise intervention is applied in the acute to step-down phases, which are the periods most critical for frailty reversal. Current dietary interventions do not address the special nutritional needs of acute cardiovascular conditions like heart failure, and may paradoxically induce a syndrome of cardiac cachexia that contributes to the downward spiral of frailty.

STUDY DESIGN:

This will be a prospective randomized clinical trial.

The investigators' proposal is a five-year study comprising of first phase (first 2-2.5 years) and second phase (next 2-2.5 years). In the first phase cardiac frail participants (up to N=500) from each healthcare transition (inpatient hospital, step-down community hospital, outpatient clinic/community) will be randomized to receive Intervention Sets or usual care. The second phase will scale up these programs. At enrolment, pre-defined study time points and end of study, participants will undergo assessments of clinical status, frailty status, cardiovascular function, nutrition, quality of life (QOL), diet/exercise behaviour, and biospecimen sampling. Three Intervention Sets will be implemented in the outpatient, step-down community hospital, and acute hospital settings. Diet intervention comprises meal sets prepared with nutrients involved in energy metabolism. During the trial, exercise intervention is performed in hospitals and community hospitals by physiotherapists. Associated factors such as dietary, comorbidities and other related habits will be tracked simultaneously during the trial

Intervention Set A: exercise sessions and meals over approximately 12 weeks. Intervention Set B : exercise sessions and meals over approximately 3 weeks. Intervention Set C: meals over approximately 3 weeks.

PROCEDURES

1. Baseline Procedures i. Cardiovascular measurements

   * Non-invasive brachial blood pressure machine
   * Echocardiography
   * Electrocardiography ii. Biospecimen collection iii. Six-minute walk test iv. Musculoskeletal Analysis v. Cardiopulmonary exercise test (CPET)/ Treadmill vi. Questionnaires vii. Timed up and go (TUG) test
2. Post-intervention procedures i. Cardiovascular measurements

   * Non-invasive brachial blood pressure machine
   * Echocardiography
   * Electrocardiography ii. Biospecimen collection iii. Six-minute walk test iv. Musculoskeletal Analysis v. Questionnaires vi. Timed up and go (TUG) test
3. Closing questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years old
* Outdoor ambulant

Exclusion Criteria:

1. Bed-bound
2. Dementia (Stage 6 onwards)
3. Residing in sheltered or nursing home
4. Cancer (to avoid confounding with cardiac disease sequelae from cancer)
5. Participation in ongoing clinical trials that involve interventional drugs or devices
6. Uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥90mmHg) despite being on treatment for hypertension
7. Low blood pressure (systolic blood pressure <90mmHg or diastolic blood pressure <40mmHg)
8. Uncontrolled atrial fibrillation (controlled atrial fibrillation is allowed)
9. Ventricular arrhythmias (such as ventricular tachycardia)
10. Renal failure on dialysis
11. Chronic kidney disease Stage 4 and above
12. Nephrotic syndrome
13. Liver cirrhosis Child's B and above
14. Inflammatory Bowel Disease
15. Severe uncontrolled gout
16. Poorly controlled Diabetes Hba1c ≥9%
17. On warfarin
18. Presence of food allergies (such as shell-fish, prawn)
19. Patient's life expectancy is expected to be less than one year at the time of potential enrolment as assessed by the investigator
20. Nasogastric or parenteral nutrition
21. Hypertrophic cardiomyopathy
22. Cardiac amyloidosis
23. Cardiac sarcoidosis

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2028-06-21 (Estimated); Study Completion 2028-06-21 (Estimated)

PRIMARY OUTCOMES:
Improvement in cardiovascular markers | at 14 weeks from baseline
  * Change in cardiovascular variables are diastolic function variables such as mitral annular velocities (m/s) OR;
  * Change in Aerobic capacity (V02, ml/kg/min)
Improvement in skeletal muscle | at 14 weeks from baseline
  Change in skeletal muscle mass (grams)
Improvement in Fried Frailty Phenotype Score (improvement in any domain) (i.e., reduction in score) | at six months from baseline

SECONDARY OUTCOMES:
Improvement in metabolite level | Three months and six months from baseline
  Any change in metabolite (microM)
Improvement in Quality of life (QOL): EuroQOL-5D-5L (higher score) | Three months and six months from baseline
  A unit increase (i.e., improvement) in QOL score

OTHER OUTCOMES:
Proportion of participants who experience a major adverse cardiovascular events | Thirty-six (36) months from baseline
  Include cardiac mortality, acute myocardial infarction, unstable angina, any revascularization, heart failure, atrial fibrillation, strokes
Other events include proportion of participants who experience : death, falls, fractures, hospitalization for any cause, admission into nursing home | Thirty-six (36) months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Angela Su-Mei Koh, MBBS, MPH, Principal Investigator — National Heart Centre Singapore
Locations (6):
- Singapore (6):
  - Alexandra Hospital, Singapore
  - National Heart Centre Singapore, Singapore
  - Changi General Hospital, Singapore
  - Sengkang General Hospital, Singapore
  - Jurong Community Hospital, Singapore
  - NHG Polyclinics, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koh AS, Gao F, Leng S, Kovalik JP, Zhao X, Tan RS, Fridianto KT, Ching J, Chua SJ, Yuan JM, Koh WP, Zhong L. Dissecting Clinical and Metabolomics Associations of Left Atrial Phasic Function by Cardiac Magnetic Resonance Feature Tracking. Sci Rep. 2018 May 25;8(1):8138. doi: 10.1038/s41598-018-26456-8. PMID 29802321
- [Background] Koh AS, Gao F, Liu J, Fridianto KT, Ching J, Tan RS, Wong JI, Chua SJ, Leng S, Zhong L, Keng BM, Huang FQ, Yuan JM, Koh WP, Kovalik JP. Metabolomic profile of arterial stiffness in aged adults. Diab Vasc Dis Res. 2018 Jan;15(1):74-80. doi: 10.1177/1479164117733627. Epub 2017 Oct 4. PMID 28976207
- [Background] Keng BMH, Gao F, Teo LLY, Lim WS, Tan RS, Ruan W, Ewe SH, Koh WP, Koh AS. Associations between Skeletal Muscle and Myocardium in Aging: A Syndrome of "Cardio-Sarcopenia"? J Am Geriatr Soc. 2019 Dec;67(12):2568-2573. doi: 10.1111/jgs.16132. Epub 2019 Aug 16. PMID 31418823
- [Background] Koh AS, Gao F, Tan RS, Zhong L, Leng S, Zhao X, Fridianto KT, Ching J, Lee SY, Keng BMH, Yeo TJ, Tan SY, Tan HC, Lim CT, Koh WP, Kovalik JP. Metabolomic correlates of aerobic capacity among elderly adults. Clin Cardiol. 2018 Oct;41(10):1300-1307. doi: 10.1002/clc.23016. PMID 30350416